CLINICAL TRIAL: NCT01899508
Title: Virtual Reality for Osteoarthritis Knee Pain Pilot
Acronym: VROA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study has been terminated, due to technically difficulties.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00045175
Record Dates: First submitted 2013-06-26; First posted 2013-07-15 (Estimated); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pain Coping Training with 3D viewer (Experimental): All participants will receive a 1 and a half hour pain coping training while using the virtual reality viewer. We are testing the feasability of using the 3D viewer in collaboration with Pain Coping training to see if people who suffer from Osteoarthritis of the knee experience some pain relief.
  Interventions: Procedure: Virtual Reality Training Session; Device: 3D viewer with iPod Touch/iPhone (or similar smartphone)

INTERVENTIONS:
Procedure: Virtual Reality Training Session — The participant will meet with an interventionist for an hour and a half long session. During this session OA knee pain will be assessed (using self report questionnaires) prior to and post a 10 minute session using the 3D viewer and having a brief pain coping skills training.
Device: 3D viewer with iPod Touch/iPhone (or similar smartphone) — The participant will meet with an interventionist for an hour and a half long session. During this session OA knee pain will be assessed (using self report questionnaires) prior to and post a 10 minute session using the 3D viewer and having a brief pain coping skills training.

SUMMARY:
This study is looking at whether virtual reality combined with pain coping skills training helps reduce pain in people who suffer from OA of the knee. Eligible participants will be asked to come into the study offices for one visit where they will fill out a couple of questionnaires, do some low impact performance tasks and be taught pain coping skills while looking into a 3D virtual reality viewer.

DETAILED DESCRIPTION:
The primary objective of this study is to examine the feasibility and acceptability of a new virtual reality (VR) protocol that uses an iPod Touch/iPhone (or similar smartphone) to deliver virtual reality (VR). The secondary objective of this study is to gather preliminary data on the efficacy and potential benefits of the VR protocol for individuals suffering from persistent osteoarthritis (OA) pain of the knees.

Study activities and population group:30 patients with a clinical diagnosis of osteoarthritis (OA) of the knee(s) will be recruited from the clinics of the Duke Division of Rheumatology and Duke Department of Orthopedic Surgery. All participants will complete screening measures, a baseline set of measures, a virtual reality training session, and post-training measures. Participants will include 30 OA patients. Inclusion criteria include: 1) having a diagnosis of OA of the knee(s), 2) age 18 or over, 3) able to read and speak English, 4) having OA related pain upon movement. 5) Self-reported normal or corrected to normal vision, 6) Self-reported normal hearing.

Cybersickness is a possible risk, a type of motion sicknesses often involving feelings of nausea, eyestrain and/or dizziness. Anticipated risks associated with cybersickness are comparable to typical "everyday" use of computers. If the participant begins to feel any effect of this type, he/she may immediately remove the virtual reality device from his/her eyes and stop the treatment. Patients will be asked to report these symptoms and will have the option of discontinuing participation if these symptoms are problematic. Third, participants may experience anxiety or distress due to questioning about thoughts, feelings, and/or their experience with OA pain. Again, participants will have the option to discontinue participation if they experience such problems in completing the measures. Finally, there is also the possibility of a breach of confidentiality. The informed consent process will address this possibility. All efforts will be made for confidentiality to be maintained. In terms of data analysis, a series of analyses will be performed to derive treatment effect size estimates (using eta squared) and their 95% confidence intervals for all outcomes. While the investigator expects mostly moderate effect sizes, given the sample size and the fact that this is a preliminary pilot study, the study team will examine within-group differences at an alpha of .10. To evaluate treatment effects on the outcome measures, the analytic strategy involves two analyses. In the first analysis, a multivariate analysis-of-variance model will be used to make within group comparisons that are unadjusted for baseline variables. In the second (primary) analysis, a multivariate analysis-of-covariance model will be used; covariates will be the pre-treatment scores on each of the outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18-85 years old
* Have a clinical diagnosis of OA of the knee
* Be able to read and write English

Exclusion Criteria:

* Can't have rheumatoid arthritis, fibromyalgia, or other chronic pain condition.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-08-17 (Actual); Study Completion 2015-08-17 (Actual)

PRIMARY OUTCOMES:
Feasibility of Virtual Reality in Pain Coping | 1.5 hours
  The primary objective of this study is to examine the feasibility and acceptability of a new virtual reality (VR) protocol that uses an iPod Touch/iPhone (or similar smartphone) to deliver virtual reality (VR). Feasibility will be assessed by examining overall accrual, attrition, and adherence to the study protocol. Ratings on a standardized measure of treatment credibility will be examined as well as a Treatment Attitude Questionnaire to assess acceptability.

SECONDARY OUTCOMES:
Change in self reported pain | 1.5 hours
  Prior to and immediately following the participant's use of the 3D viewer they will be asked to rate their pain and complete questionnaires using the following scale to rate pain:
  Pain Self-Efficacy. Self-efficacy will be measured using the self-efficacy for pain management subscale of the 22-item Chronic Pain Self-Efficacy Scale (CPSS). The pain management subscale consists of 5 questions measuring levels of self-efficacy for pain management. For example, "How certain are you that you can decrease your pain quite a bit?", "How certain are you that you can continue most of your daily activities?" and "How certain are you that you can keep your pain from interfering with your sleep?". Participants circle the number that best corresponds with their certainty on a 10-point scale ranging in 10-point increments from 10 (very uncertain) to 100 (very certain). Scores for each question are averaged to give an overall value for self-efficacy for pain management.

CONTACTS AND LOCATIONS:
Overall Officials: Franicis Keefe, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center department Psychiatry, Durham, North Carolina, United States